CLINICAL TRIAL: NCT04455763
Title: Autologous Stromal Vascular Fraction in the Treatment of Thumb Basal Joint Osteoarthritis - ReMeDY SVF -Trial
Brief Title: Autologous Stromal Vascular Fraction in the Treatment of Thumb Basal Joint Osteoarthritis
Acronym: REMEDY SVF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Töölö Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Samuli Aspinen, Principal investigator, Töölö Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1866/2020
Record Dates: First submitted 2020-06-28; First posted 2020-07-02 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Thumb Osteoarthritis
Keywords: Thumb Osteoarthrosis; Stromal Vascular Fraction
MeSH Terms: interventions — Splints

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SVF (Experimental): Thumb carpometacarpal injection with adipose-derived SVF combined with splinting
  Interventions: Procedure: SVF; Other: Splint
- Splint (Active Comparator): Thumb carpometacarpal osteoarthrosis treated with splinting only
  Interventions: Other: Splint

INTERVENTIONS:
Procedure: SVF — Adipose-derived stromal vascular fraction
  Arms: SVF
Other: Splint — Thumb brace (Actimove® Rhizo Forte)

SUMMARY:
Trial purpose is to research the outcome after thumb carpometacarpal injection with stromal vascular fraction (SVF) derived from adipose tissue. The study compares SVF injection therapy with thumb splinting vs. splinting only.

Patients with radiologically and clinically confirmed Eaton-Glickel II osteoarthritis are randomized (1:1 computer generated sequence with random block size) to two parallel groups and will undergo SVF injection and splinting vs. splinting only.

Baseline data is collected preoperatively and patients are followed at 1, 3 and 6 months after enrollment. The primary end-point is 6 months and the primary outcome is pain visual analogue scale and patient-rated wrist evaluation (PRWE).

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Eaton-Glickel II thumb CMC osteoarthrosis
* Symptom duration > 3 months
* Pain visual analogue score > 30 mm
* < 3 months of treatment with thumb splinting
* American Society of Anaesthesiologists physical status (ASA) I-III
* Fluent in written and spoken Finnish

Exclusion Criteria:

* Age <40 or >70 years
* Eaton-Glickel I, III-IV
* Symptom duration < 3 months
* Pain VAS < 30 mm
* Post-traumatic osteoarthrosis of thumb CMC I
* Rheumatoid arthritis or other inflammatory joint disease
* The use of per oral corticosteroids or other immunomodulatory drugs
* Less than 6 months after another operation of the same upper limb
* Other condition of the same upper limb requiring surgery
* Malnutrition
* Neurological condition affecting upper limb function
* Heavy smoking (> 20 cigarettes per day)
* Alcohol or drug abuse
* Previous history or active cancer
* Previous history of allergic reaction to local anaesthetic

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Pain (Visual Analogue Scale) | 6 months
  The VAS is derived by health care professional question of pain in scale 0 to 100 mm (0 mm =no pain, 100 mm =worst possible pain)
Patient-Rated Wrist Evaluation (PRWE) | 6 months
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists two subscales: Pain and Function (0=best possible outcome, 10=worst possible outcome)

SECONDARY OUTCOMES:
Global improvement | 6 months
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better
Grip strength | 6 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side
Key pinch strength | 6 months
  Key pinch strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side
Michigan Hand Outcomes Questionnaire (MHQ) | 6 months
  The MHQ comprises of 37 core questions to measure hand-specific outcomes containing six distinct scales: overall hand function, activities of daily living, pain, work performance, aesthetics and patient satisfaction with hand function.
Complications | 6 months
  Incidence of complications (hemaetoma, injection site infection etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Samuli Aspinen, M.D., Ph.D., Principal Investigator — HUS Töölö Hospital
Locations (1):
- Töölö Hospital (Helsinki University Hospital), Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No